CLINICAL TRIAL: NCT00101374
Title: A Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Effect of Leflunomide on HIV-1 Associated Immune Proliferation In Vivo
Brief Title: Effect of Leflunomide on T Cell Proliferation in HIV-Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050065; 05-I-0065
Record Dates: First submitted 2005-01-07; First posted 2005-01-10 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-02-02

CONDITIONS: HIV Infections
Keywords: Immunomodulatory Drug; Antiviral; Ki67+; Immune Activation; T Cell Proliferation; HIV; Activated CD4+T-cell; Proliferation
MeSH Terms: conditions — HIV Infections | interventions — Leflunomide

INTERVENTIONS:
Drug: Leflunomide

SUMMARY:
This study will evaluate the effect of leflunomide on the life cycle of a specific immune cell called CD4+ T cell in HIV-infected patients. Leflunomide is approved by the Food and Drug Administration for treating rheumatoid arthritis. It works by blocking cell division in activated T cells. In HIV infection, the HIV virus causes increased activation of T cells. The activated cells become infected and die. Activation may also cause the death of T cells that are not infected with HIV. T cells are necessary for the body to fight infections and cancer. This study will see if leflunomide can block T-cell division and possibly reduce the number of cells that die, reduce the number of cells in which HIV can reproduce, and lead to a lower level of HIV virus in the body.

HIV-infected patients between 18 and 65 years of age who have 1) HIV viral levels of 1,000 copies/mL or more, 2) a CD4+ T-cell count of 350 cells/mm3 or more, and 3) a CD4+ T-cell count that has never been less than 200 cells/mm3 may be eligible for this study. Candidates are screened with a medical history, physical examination, blood and urine tests, chest x-ray, and electrocardiogram (EKG).

Participants are randomly assigned to take leflunomide or placebo (a substance with no active ingredient) every day for 28 days. They come to the clinic three times during the first 29 days of the study (days 1, 15, and 29) for a physical examination and review of any drug side effects. Patients taking placebo end their participation on day 29. Patients taking leflunomide stop taking the drug on day 29 and begin taking cholestyramine three times a day for 11 days out of the next 14 days to clear the leflunomide from their body. On day 43, they return to the clinic to have their leflunomide level checked to make sure that only very little or none of the drug remains in the body. If the level is low, patients end their participation on or around day 57. If the level remains high, they repeat the cholestyramine treatment.

DETAILED DESCRIPTION:
Increased T cell turnover is one of the main abnormalities observed in HIV infected patients and one of the main mechanisms leading to CD4 lymphopenia. This has led to the hypothesis that medications that act directly to suppress immune activation and normalize T cell turnover, could be used in HIV infection. The purpose of this protocol is to evaluate the effect of the immunomodulatory agent, leflunomide, on CD4+ T cell proliferation in HIV infected adults. HIV infected adults who have stable HIV viral loads and are not taking antiretrovirals will receive leflunomide or placebo for 28 days. CD4+ T cell proliferation will be measured as percent Ki67 expression, and the change in expression from baseline to day 28 will be compared between groups. Various studies measuring immune parameters such as CD4+ and CD8+ T cells counts and level of activation will be collected as well as safety studies and HIV viral loads. The primary study risk is adverse reaction to leflunomide. The study will be double-blinded randomized 2:1 (leflunomide versus placebo) and will be reviewed by a DSMB. Total enrollment for the study will be 18 patients.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age greater than or equal 18 and less than or equal to 65 years.
* HIV infected.
* CD4+ cell count greater than or equal to 350 cells/mm(3) at screening and historical nadir (since diagnosis of HIV) of greater than or equal to 200 cells/mm(3).
* Plasma HIV viral load greater than or equal to 1,000 copies/mL at screening.
* Ability to understand and sign informed consent and willingness to comply with the study requirements and clinic policies.
* Must have a primary care physician who will be taking care of patients for their HIV infection.
* Female study subjects of reproductive potential (defined as girls who have reached menarche or women who have not been post-menopausal for at least 24 consecutive months, i.e., who have had menses within the preceding 24 months or have not undergone a sterilization procedure (hysterectomy or bilateral oophorectomy), must have a negative serum or urine pregnancy test.
* Agreement not to participate in a conception process (eg. active attempt to become pregnant or impregnate, sperm donation, or in vitro fertilization) and to follow strict contraceptive measures while on study.
* If participating in sexual activity that could lead to pregnancy, the study volunteer must agree that two reliable methods of contraception will be used simultaneously during the entire study. Acceptable forms of contraception include:

Condoms (male or female) with or without a spermicidal agent. Condoms are recommended because their appropriate use is the only contraception method effective for preventing HIV transmission.

Diaphragm or cervical cap with spermicide.

IUD.

Hormonal-based contraception.

Study subjects who are not of reproductive potential (women who have been post-menopausal for at least 24 consecutive months, women who have undergone hysterectomy or bilateral oophorectomy, or prepubescent boys or men who have documented azoospermia) are eligible without requiring the use of contraception.

Written or oral documentation communicated by clinician or clinician's staff of one of the following:

Physician report/letter.

Operative report or other source documentation in the patient record (a laboratory report of azoospermia is required to document successful vasectomy).

Discharge summary.

Laboratory report of azoospermia.

FSH measurement elevated into the menopausal range as established by the reporting laboratory.

EXCLUSION CRITERIA:

* Current treatment with antiretrovirals or use of antiretrovirals within 12 weeks of screening.
* Intention of start antiretroviral regimen within 64 day study period.
* Previous treatment with leflunomide.
* Previous treatment with IL-2.
* Treatment with immunomodulatory agents (including hydroxyurea, mycophenolate, cyclosporine, rapamycin, anti-HIV vaccines, interleukins other than IL-2, interferons) within 60 days of study.
* Treatment with systemic corticosteroids within 30 days of study.
* Inability or unwillingness to discontinue drugs (except NSAIDS) that are metabolized by P450 2C9 isoenzyme (see Appendix A- Medications Metabolized by CYP 2C9 and Contraindicated During Treatment Period).
* Inability or unwillingness to discontinue hepatotoxic drugs (eg. isoniazid, rifampin, HMG CoA reductase inhibitors).
* Inability or unwillingness to discontinue drug that interact with cholestyramine (eg. have diminished absorption with cholestyramine) (see Appendix B- Medications that have Interactions with Cholestyramine).
* Current use of or known intolerance of cholestyramine or bile acid sequestering resins.
* History of familial hyperlipoproteinemia type III, IV or V.
* Active bacterial infection within 4 weeks of screening.
* History of AIDS-defining illness (category C) (see Appendix C - CDC AIDS Classification Criteria).
* Hepatitis B or C infection.
* Acute or chronic liver disease from any cause (eg. alcoholic hepatitis or alcohol induced cirrhosis, autoimmune hepatitis, primary biliary cirrhosis, sclerosing cholangitis, Wilson's disease, hemochromatosis) which the investigator feels would compromise the subject's safety.
* History of biliary obstruction.
* Current alcohol abuse or unwillingness to abstain from alcohol use for study period.
* History of hypertension that is not controlled (less than 140/80 mm/Hg) on a single antihypertensive agent.
* Abnormal laboratory findings: hemoglobin less than 10 g/dL; ANC less than 1000/mm(3); platelets less than 100,000/mm(3); creatine above the upper limit of normal; ALT or alkaline phosphatase greater than 1.25 times the upper limit of normal; AST greater than 1.25 times the upper limit of normal (subjects with isolated AST elevation, higher than normal CPK values in the absence of liver disease and compatible history such as intense exercise will be allowed to re-screen if the study investigators suspect that the elevated AST is of muscular origin) direct bilirubin greater than 1.5 times the upper limit of normal; total bilirubin greater than 2 times the upper limit of normal lipase greater than 1.5 times the upper limit of normal; PT greater than 1.1 times the upper limit of normal; PTT greater than 1.5 times the upper limit of normal.
* History of malignant neoplasm except in situ anogenital carcinoma, adequately treated basal or squamous cell carcinoma of the skin or solid tumors treated with curative therapy and disease free for at least five years.
* Significant medical or psychiatric disorder which the investigator feels would interfere with the subject's ability to participate or would compromise safety.
* Women who are currently pregnant or breast-feeding.
* History of interstitial lung disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2005-01-05; Primary Completion 2008-05-21 (Actual); Study Completion 2008-05-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Grossman Z, Meier-Schellersheim M, Sousa AE, Victorino RM, Paul WE. CD4+ T-cell depletion in HIV infection: are we closer to understanding the cause? Nat Med. 2002 Apr;8(4):319-23. doi: 10.1038/nm0402-319. No abstract available. PMID 11927927
- [Background] McCune JM. The dynamics of CD4+ T-cell depletion in HIV disease. Nature. 2001 Apr 19;410(6831):974-9. doi: 10.1038/35073648. PMID 11309627
- [Background] Sousa AE, Carneiro J, Meier-Schellersheim M, Grossman Z, Victorino RM. CD4 T cell depletion is linked directly to immune activation in the pathogenesis of HIV-1 and HIV-2 but only indirectly to the viral load. J Immunol. 2002 Sep 15;169(6):3400-6. doi: 10.4049/jimmunol.169.6.3400. PMID 12218162
- [Derived] Read SW, DeGrezia M, Ciccone EJ, DerSimonian R, Higgins J, Adelsberger JW, Starling JM, Rehm C, Sereti I. The effect of leflunomide on cycling and activation of T-cells in HIV-1-infected participants. PLoS One. 2010 Aug 3;5(8):e11937. doi: 10.1371/journal.pone.0011937. PMID 20689824